CLINICAL TRIAL: NCT04896281
Title: Phenylalanine-free Diet Lowers the Blood Phenylalanine Levels in Patients With High Phenylalanine Level in the Intensive Care Unit
Brief Title: Phenylalanine-free Diet for Patients With Secondary Hyperphenylalaninemia in ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202100028A3
Record Dates: First submitted 2021-04-26; First posted 2021-05-21 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Non-Phenylketonuric Hyperphenylalaninemia
Keywords: phenylalanine; intensive care unit; nutritional intervention
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- phenylalanine-free diet (Experimental): phenylalanine-free diet for patients with hyperphenylalaninemia
  Interventions: Dietary Supplement: Phenylalanine-free milk

INTERVENTIONS:
Dietary Supplement: Phenylalanine-free milk — Once a plasma PHE level of ≥ 95 μM is noted, phenylalanine-free diet (Phenex-2®, Abbott Nutrition, Ohio, USA; or Phenyl-Free 2®, Mead Johnson Nutrition, Minnesota, USA) is started as the only nutrition source for enteral feeding, as per the recommendation of dieticians, in the following 4 days. The phenylalanine-free diet is free of PHE but is enriched with protein, potassium, tyrosine, and antioxidant micronutrients. After the completion of the study, diet will be back to normal diet for all patients.

SUMMARY:
Hyperphenylalaninemia is not only present in patients with congenital phenylketonuria. In adults with critical illness, hyperphenylalaninemia is noted in some patients and is associated with high mortality rate. Hyperphenylalaninemia can cause metabolic acidosis, brain dysfunction, and metabolic disturbance. The investigators would like to see whether the phenylalanine-free milk for congenital phenylketonuria is also effective in lowering the blood phenylalanine concentrations in patients with critical illness in intensive care unit and hyperphenylalaninemia.

DETAILED DESCRIPTION:
Background:

Patients in the intensive care unit often suffer from problems such as high metabolic rate and high tissue breakdown rate under the severe stress of critical diseases. Phenylalanine is an amino acid in the human body and is rich in muscle tissue. However, current studies have found that if the concentration of phenylalanine in the blood is abnormally increased, it may indicate that the tissue is decomposing in large quantities. This phenomenon may be related to disease severity. Our recent observational study of patients in the intensive care unit (ICU) found that patients with elevated blood phenylalanine had a four-fold increase in mortality within one year.

The most common cause of phenylalanine concentration elevation in the blood is a rare disease that occurs in infants with congenital metabolic abnormalities, called congenital phenylketonuria (PKU). The abnormally elevated phenylalanine concentration can lead to toxicity and cause brain hypoplasia, mental retardation, consciousness disturbance, and even seizure. These PKU patients must be treated with milk diet that contains low amount of phenylalanine in order to lower the phenylalanine concentrations. At present, in medicine, although there have been clear medical care strategy for infants with congenital PKU, there is still no clear medical care strategy for adult patients.

Research purpose: To investigate whether patients with high blood phenylalanine concentration in the intensive care unit can reduce the blood phenylalanine concentration by a diet without phenylalanine, so as to develop personalized high-quality and specific treatments.

Methods:

The investigators aim to have complete study in 70 patients (based on our previous study, to recruit 70 patients with high phenylalanine, the investigators need 300 ICU patients for screening).

Intervention protocol:

Once a plasma phenylalanine level of ≥ 95 μM is noted, phenylalanine-free diet (Phenex-2®, Abbott Nutrition, Ohio, USA; or Phenyl-Free 2®, Mead Johnson Nutrition, Minnesota, USA) is started as the only nutrition source for enteral feeding, as per the recommendation of dieticians, in the following 4 days. The phenylalanine-free diet is free of phenylalanine but is enriched with protein, potassium, tyrosine, and antioxidant micronutrients. After the completion of the study, diet will be back to normal diet for all patients.

Study end points: the 5-day study period completed.

Blood sampling and examination for Phenylalanine measurement (dry blood spot) Fasting phenylalanine level will be measured by LC/MS-MS using the dry blood spot method (blood sample is collected by finger sting) in all included patients in the next morning after informed consent signed. Blood applied on filter cards is dried for at least 3 h at room temperature. Dry blood spot cards are stored at room temperature for 0-6 days prior to analyses. Phenylalanine concentrations in dry blood spot are measured with LC-MS/MS, using a calibration curve in 0.1 N HCl. The report will be received one day after dry blood spot collected. Once the result of measurement shows the concentration of phenylalanine ≥95 μM, this patient is enrolled for formal study. All enrolled patients will take the measurement of phenylalanine levels by dry blood spot every 12 hours for the following 4 days until study protocol finished.

Phenylalanine measurement by UPLC:

In the meanwhile, fasting blood will be collected by venipuncture in EDTA-containing tubes on the morning of screening, 2 and 4 days after diet intervention. The collected blood will be used to measure phenylalanine level by UPLC (ultra-performance liquid chromatography). Plasma samples (100μL) are precipitated with 10% sulfosalicylic acid. After protein precipitation and centrifugation, derivatization is initiated by AQC in acetonitrile. Amino acids are then analyzed using the ACQUITY UPLC System, consisting of a Binary Solvent Manager, a Sample Manager, and a Tunable UV detector. The investigators use EmpowerTM 2 Software to control the system and collect data. Separations are performed on a 2.1×100mm ACQUITY BEH C18 column at a flow rate of 0.70mL/min. The average intra-assay coefficient of variation is 2.6% for phenylalanine. The total coefficient of variation is 2.7% for phenylalanine. The detection limit is 3.3μM for phenylalanine. The linear range is 25-500 μM.

APACHE II scores Disease severity is evaluated by calculating APACHE II score on the first day of ICU admission.

ELIGIBILITY:
Inclusion Criteria:

1. had Acute Physiology And Chronic Health Evaluation (APACHE II) scores of ≥15;
2. were expected to stay in the ICU >48 hours;
3. patients with baseline PHE levels of ≥95 uM;
4. were over 20 years old.

Exclusion Criteria:

1. patients with comorbid disorders other than the main cause for admission that might compromise their survival within three months, such as terminal stage cancer;
2. patients with expected survival <3 days.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
fasting plasma phenylalanine concentration | Baseline to day 5
  fasting plasma phenylalanine concentration at baseline and at the end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: CHAO-HUNG WANG, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital, Keelung
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No
undecided